CLINICAL TRIAL: NCT01480076
Title: An Open-Label, Multicenter, Multinational Study to Assess the Effect of Long-Term Prolonged-Release Fampridine (BIIB041) 10 mg Twice Daily on Quality of Life as Reported by Subjects With Multiple Sclerosis
Brief Title: Open-Label Study to Assess the Effect of Long-Term Prolonged-Release Fampridine (BIIB041) on Quality of Life as Reported by Participants With Multiple Sclerosis
Acronym: ENABLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218MS403
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Quality of Life; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

ARMS (1):
- (BIIB041) Fampridine (Experimental): All participants take 10 mg fampridine twice daily for the first 4 weeks. If deemed a treatment responder, a participant continues 10 mg fampridine twice daily for 44 weeks. Treatment non-responders can continue without treatment by completing quality of life questionnaires.
  Interventions: Drug: Fampridine

INTERVENTIONS:
Drug: Fampridine — Supplied as a 10 mg twice daily tablet and taken twice daily. Doses must be spaced at least 12 hours apart.
  Other Names: Fampyra; BIIB041; Ampyra; dalfampridine; fampridine prolonged-release tablets

SUMMARY:
The primary objective of the study is to assess the effect of long-term treatment with prolonged-release fampridine (BIIB041) 10 mg twice daily on the physical component scale (PCS) of the Short Form 36 Health Status Questionnaire (SF-36) as reported by treatment responders. The secondary objectives of this study are to compare the change in the PCS of the SF-36 between treatment responders and non-responders, to evaluate change from baseline in additional quality of life measures among treatment responders as well as changes from baseline in treatment responders versus non-responders and to assess the safety and tolerability of prolonged-release fampridine 10 mg twice daily.

DETAILED DESCRIPTION:
This study has 2 components: a 4-week run-in period during which participants are treated with prolonged-release fampridine and undergo subjective and objective assessments of walking ability, the results of which are used to determine who responded to study treatment, and an observational period, during which treatment responders will continue prolonged-release fampridine treatment. The participants who do not meet the criteria to continue study treatment will be offered the opportunity to continue study participation but will not continue prolonged-release fampridine treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local subject privacy regulations.
* Must have a diagnosis of primary-progressive, secondary-progressive, progressive-remitting, or relapsing-remitting multiple sclerosis (MS) per revised McDonald Committee criteria ([Polman et al, 2011]) as defined by Lublin and Reingold [Lublin and Reingold 1996] of at least 3 months duration.
* Have a walking impairment as determined by the Investigator.
* Able to perform the Timed 25-foot Walk Test with or without a walking aid.
* Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.
* Able to understand and comply with the requirements of the protocol.

Key Exclusion Criteria:

* Known allergy to pyridine-containing substances or to any of the inactive ingredients in the prolonged-release fampridine tablet.
* Any history of seizure, epilepsy, or other convulsive disorder, with the exception of febrile seizures in childhood.
* An estimated creatinine clearance of <80 mL/minute.
* Subject needs to take medicinal products that are inhibitors of organic cation transporter 2 (OCT2 [e.g., cimetidine]).
* Female subjects who are currently pregnant or who are considering becoming pregnant while participating in the study.
* Female subjects who are currently breastfeeding.
* Previous exposure to fampridine.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (59):
- Australia (9):
  - Research Site, Concord, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research Site, Box Hill, Victoria
  - Research Site, Clayton, Victoria
  - Research Site, Fitzroy, Victoria
  - Research Site, Heidelberg, Victoria
- Belgium (10):
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Diepenbeek
  - Research Site, Fraiture-en-Condroz
  - Research Site, Ghent
  - Research Site, Liège
  - Research Site, Melsbroek
  - Research Site, Overpelt
  - Research Site, Sijsele-Damme
  - Research Site, Wilrijk
- Research Site, Copenhagen, Denmark
- France (11):
  - Research Site, Nice, Alpes-Maritimes
  - Research Site, Strasbourg, Bas-Rhin
  - Research Site, Caen, Calvados
  - Research Site, Bordeaux, Gironde 5
  - Research Site, Rennes, Ille-et-Vilaine
  - Research Site, Nantes, Loire-Atlantique 6
  - Research Site, Reims, Marne
  - Research Site, Clemont-Ferrand, Rhone
  - Research Site, Paris, Seine-Saint-Denis 14
  - Research Site, Amiens, Somme
  - Research Site, Paris
- Germany (10):
  - Research Site, Heidenheim, Bad Wuerttemberg
  - Research Site, Kassel, Hesse
  - Research Site, Oldenburg, Lower Saxony
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Berlin
  - Research Site, Erbach im Odenwald
  - Research Site, Hamburg
  - Research Site, Jena
  - Research Site, Osnabrück
  - Research Site, Schwendi
- Italy (5):
  - Research Site, Bari
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
- Netherlands (4):
  - Research Site, Eindhoven
  - Research Site, Hoorn
  - Research Site, Nijmegen
  - Research Site, Tilburg
- Portugal (4):
  - Research Site, Amadora
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
- United Kingdom (5):
  - Research Site, Salford, Greater Manchester
  - Research Site, Nottingham, Northamptonshire
  - Research Site, Glasgow, Stirlingshire
  - Research Site, Liverpool
  - Research Site, London

REFERENCES:
- [Background] Macdonell R, Nagels G, Laplaud DA, Pozzilli C, de Jong B, Martins da Silva A, Nicholas R, Lechner-Scott J, Gaebler JA, Agarwal S, Wang P, Yeh M, Hovenden M, Soelberg Sorensen P. Improved patient-reported health impact of multiple sclerosis: The ENABLE study of PR-fampridine. Mult Scler. 2016 Jun;22(7):944-54. doi: 10.1177/1352458515606809. Epub 2015 Oct 7. PMID 26447066

RESULTS

PARTICIPANT FLOW:
Groups:
- Fampridine: All participants took 10 mg fampridine twice daily for the first 4 weeks. If deemed a treatment responder, the participant continued 10 mg fampridine twice daily for 44 weeks. Treatment non-responders continued without treatment by completing quality of life questionnaires.
Period: Overall Study
Arm/Group | Fampridine
Started | 901 (enrolled and started run-in treatment)
Intent to Treat Population | 835 (Received ≥1 dose of study drug & provided ≥1 efficacy assessment at Baseline & the 3-month visit.)
Completed | 611
Not Completed | 290
Not completed — Run-in Failure | 52
Not completed — Adverse Event | 39
Not completed — Death | 2
Not completed — Disease Progression | 5
Not completed — Non-compliance With Study Protocol | 15
Not completed — Withdrawal by Subject | 105
Not completed — Lost to Follow-up | 7
Not completed — Investigator Decision | 13
Not completed — Other | 52

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: all participants who received at least 1 dose of study treatment and who provided at least 1 efficacy assessment at Baseline and the 3-month visit.
Groups:
- Responder: Participants took 10 mg fampridine twice daily for the first 4 weeks. If deemed a treatment responder, the participant continued 10 mg fampridine twice daily for 44 weeks.
- Non-responder: Participants took 10 mg fampridine twice daily for the first 4 weeks. Treatment non-responders continued without treatment by completing quality of life questionnaires.
- Total: Total of all reporting groups
Arm/Group | Responder | Non-responder | Total
Number analyzed (Participants) | 707 | 128 | 835
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (9.70) | 50.5 (10.0) | 49.5 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 402 | 79 | 481
  Male | 305 | 49 | 354

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Physical Component Scale (PCS) of the Short Form 36 Health Status Questionnaire (SF-36) At Months 3, 6, 9, and 12: Responders
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the mental component summary (MCS) score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Increases from baseline indicate improvement. Within-group least squares means are presented.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: Participants in the intent-to-treat population (all participants who received at least 1 dose of study treatment and who provided at least 1 efficacy assessment at Baseline and the 3-month visit) who were included in the mixed effect model for repeated measures analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Responder: Participants took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment responders continued 10 mg fampridine twice daily for 44 weeks.
Arm/Group | Responder
Number analyzed (Participants) | 666
units on a scale
  Month 3 | 4.2 (0.36)
  Month 6 | 3.4 (0.38)
  Month 9 | 3.2 (0.37)
  Month 12 | 2.9 (0.37)
Statistical Analysis 1: Comparison: Responder; Month 3: Mixed effect model for repeated measures with visit, baseline PCS score, baseline Expanded Disability Status Scale (EDSS) score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model — within group p-value
Statistical Analysis 2: Comparison: Responder; Month 6: Mixed effect model for repeated measures with visit, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model — within group p-value
Statistical Analysis 3: Comparison: Responder; Difference of Month 3 versus Month 6: Mixed effect model for repeated measures with visit, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0007, mixed effect model; least squares mean = 0.8, Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Responder; Month 9: Mixed effect model for repeated measures with visit, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model — within-group p-value
Statistical Analysis 5: Comparison: Responder; Difference of Month 6 versus Month 9: Mixed effect model for repeated measures with visit, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2531, mixed effect model; least squares mean = 0.2, Standard Error of Mean 0.21
Statistical Analysis 6: Comparison: Responder; Month 12: Mixed effect model for repeated measures with visit, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model — within group p-value
Statistical Analysis 7: Comparison: Responder; Difference of Month 9 versus Month 12: Mixed effect model for repeated measures with visit, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2299, mixed effect model; least squares mean = 0.3, Standard Error of Mean 0.21

2. Secondary Outcome: Change From Baseline in the PCS of the SF-36 at Months 3, 6, 9, and 12: Responders Versus Non-responders
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the MCS score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Increases from baseline indicate improvement. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12). In contrast to the primary endpoint, this analysis was done using data from both responder and non-responder groups; therefore, 'responder group' and 'visit by responder group interaction' were included as fixed effects.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Non-responder: Participants took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment non-responders continued without treatment by completing quality of life questionnaires.
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 666 | 81
units on a scale
  Overall | 3.3 (0.34) | -0.4 (0.63)
  Month 3 | 4.0 (0.36) | -0.2 (0.67)
  Month 6 | 3.3 (0.37) | 0.2 (0.77)
  Month 9 | 3.0 (0.37) | -1.1 (0.80)
  Month 12 | 2.8 (0.37) | -0.5 (0.81)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5405, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 3.7, Standard Error of Mean 0.58
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7272, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 4.3, Standard Error of Mean 0.64
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7484, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 3.0, Standard Error of Mean 0.75
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1877, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 4.1, Standard Error of Mean 0.78
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5460, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline PCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 3.3, Standard Error of Mean 0.79

3. Secondary Outcome: Change From Baseline in the MCS of the SF-36 At Months 3, 6, 9, and 12
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the MCS score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Increases from baseline indicate improvement. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 667 | 81
units on a scale
  Overall | 3.1 (0.53) | 0.1 (0.95)
  Month 3 | 4.2 (0.55) | -0.6 (1.03)
  Month 6 | 3.3 (0.56) | 0.6 (1.12)
  Month 9 | 2.3 (0.58) | 1.0 (1.22)
  Month 12 | 2.5 (0.57) | -0.6 (1.21)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9073, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0009, mixed effect model; least squares mean = 3.0, Standard Error of Mean 0.89
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5542, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 4.8, Standard Error of Mean 0.99
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5810, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0140, mixed effect model; least squares mean = 2.7, Standard Error of Mean 1.08
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4138, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2740, mixed effect model; least squares mean = 1.3, Standard Error of Mean 1.19
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6453, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MCS score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0090, mixed effect model; least squares mean = 3.1, Standard Error of Mean 1.18

4. Secondary Outcome: Change From Baseline in the Multiple Sclerosis Impact Scale (MSIS-29) Physical Score at Months 3, 6, 9, and 12
Description: The MSIS-29 is a disease specific patient-reported outcome measure that has been developed and validated to examine the physical and psychological impact of MS from a patient's perspective; it measures 20 physical items and 9 psychological items. Sum of 20 physical condition items converted into a 0-100 score range, where missing items are imputed by average of total of non-missing items when no more than 50% are missing (otherwise the total score is missing). A lower total score indicates less physically-related impact while a higher total score indicates greater physically-related impact on a participant's functioning. Decreases from Baseline indicate improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 669 | 79
units on a scale
  Overall | -10.3 (0.99) | -2.1 (1.79)
  Month 3 | -13.0 (1.00) | -2.1 (1.83)
  Month 6 | -10.6 (1.03) | -3.0 (1.99)
  Month 9 | -8.9 (1.06) | -0.3 (2.19)
  Month 12 | -8.6 (1.06) | -2.8 (2.23)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2475, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = -8.2, Standard Error of Mean 1.66
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2422, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = -10.9, Standard Error of Mean 1.72
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1262, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = -7.6, Standard Error of Mean 1.90
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8858, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = -8.6, Standard Error of Mean 2.12
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2111, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 physical score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0072, mixed effect model; least squares mean = -5.8, Standard Error of Mean 2.16

5. Secondary Outcome: Change From Baseline in MSIS-29 Psychological Score at Months 3, 6, 9, and 12
Description: The MSIS-29 is a disease specific patient-reported outcome measure that has been developed and validated to examine the physical and psychological impact of MS from a patient's perspective; it measures 20 physical items and 9 psychological items. Sum of 9 psychological condition items converted into a 0-100 score range, where missing items are imputed by average of total of non-missing items when no more than 50% are missing (otherwise the total score is missing). A lower total score indicates less psychologically-related impact while a higher total score indicates greater psychologically-related impact on a participant's functioning. Decreases from Baseline indicate improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 669 | 79
units on a scale
  Overall | -7.8 (0.97) | -1.0 (1.77)
  Month 3 | -9.6 (1.01) | -0.2 (1.91)
  Month 6 | -7.7 (1.03) | -2.6 (2.06)
  Month 9 | -6.8 (1.06) | -0.8 (2.26)
  Month 12 | -7.0 (1.06) | -0.5 (2.34)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5577, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = -6.7, Standard Error of Mean 1.64
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9365, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = -9.4, Standard Error of Mean 1.82
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2008, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0102, mixed effect model; least squares mean = -5.1, Standard Error of Mean 1.98
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7134, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0066, mixed effect model; least squares mean = -6.0, Standard Error of Mean 2.20
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8202, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder status, visit by responder status interaction, baseline MSIS-29 psychological score, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0049, mixed effect model; least squares mean = -6.4, Standard Error of Mean 2.28

6. Secondary Outcome: Change From Baseline in the Activities Limitation Scale of the Patient-Reported Indices for Multiple Sclerosis (PRIMUS) at Months 3, 6, 9, and 12
Description: The PRIMUS activity measure is a 15-item assessment of patient-reported activities of daily living. The total score was calculated as sum of all 15 items converted into a 0-30 range, where missing items were imputed by average of non-missing total when no more than 50% of items were missing (otherwise, the total score is missing). Higher score indicates worse condition. A decrease from Baseline indicates improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 498 | 45
units on a scale
  Overall | -1.4 (0.22) | 0.8 (0.56)
  Month 3 | -2.3 (0.23) | -0.4 (0.58)
  Month 6 | -1.4 (0.25) | 0.8 (0.70)
  Month 9 | -1.2 (0.25) | 1.8 (0.73)
  Month 12 | -0.8 (0.26) | 1.1 (0.83)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1324, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = -2.3, Standard Error of Mean 0.56
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4759, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0016, mixed effect model; least squares mean = -1.9, Standard Error of Mean 0.59
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2489, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0017, mixed effect model; least squares mean = -2.2, Standard Error of Mean 0.71
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0126, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = -3.1, Standard Error of Mean 0.75
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0033, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1758, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the total activity limitation score of PRIMUS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0246, mixed effect model; least squares mean = -1.9, Standard Error of Mean 0.84

7. Secondary Outcome: Change From Baseline in the Current Health State of EuroQoL Descriptive System of Health-related Quality of Life States Consisting of 5 Dimensions (EQ-5D) Visual Analog Scale (VAS) at Months 3, 6, 9, And 12
Description: EQ-5D is a participant-answered questionnaire containing a descriptive system of 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression and a VAS on health state. The EQ-5D VAS ranges from 0 (worst health state) to 100 (best health state). An increase from baseline indicates improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 659 | 79
units on a scale
  Overall | 6.7 (0.95) | -4.4 (1.73)
  Month 3 | 8.0 (1.00) | -3.2 (1.91)
  Month 6 | 6.1 (1.02) | -3.6 (2.06)
  Month 9 | 6.3 (1.04) | -4.9 (2.21)
  Month 12 | 6.3 (1.05) | -6.0 (2.34)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0111, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder Versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 11.1, Standard Error of Mean 1.61
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0970, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder Versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 11.1, Standard Error of Mean 1.82
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0789, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder Versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 9.7, Standard Error of Mean 2.00
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0284, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder Versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 11.2, Standard Error of Mean 2.16
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0108, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder Versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of the current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; least squares mean = 12.3, Standard Error of Mean 2.29

8. Secondary Outcome: Change From Baseline in the Index Scores of EQ-5D at Months 3, 6, 9, and 12
Description: EQ-5D is a participant-answered questionnaire containing a descriptive system on 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression and a VAS on health state. The scores on the 5 dimensions of descriptive system can be converted into an index score by applying United Kingdom (UK) weights. EQ-5D index score ranges from 1 to -0.59, and 1 reflects the best outcome. An increase from baseline indicates improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 661 | 78
units on a scale
  Overall | 0.05 (0.01) | 0.00 (0.02)
  Month 3 | 0.07 (0.01) | 0.01 (0.02)
  Month 6 | 0.05 (0.01) | 0.01 (0.02)
  Month 9 | 0.04 (0.01) | 0.01 (0.03)
  Month 12 | 0.04 (0.01) | -0.01 (0.03)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8392, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0162, mixed effect model; least squares mean = 0.04, Standard Error of Mean 0.02
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6956, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0042, mixed effect model; least squares mean = 0.06, Standard Error of Mean 0.02
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7949, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0679, mixed effect model; least squares mean = 0.04, Standard Error of Mean 0.02
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0027, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8053, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2638, mixed effect model; least squares mean = 0.03, Standard Error of Mean 0.03
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0007, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8502, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of current health state of EQ-5D scores, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0917, mixed effect model; least squares mean = 0.05, Standard Error of Mean 0.03

9. Secondary Outcome: Change From Baseline in Percent Work Time Missed Due to MS, by the Work Productivity and Activity Impairment-Specific Health Problem (WPAI-SHP) Questionnaire at Months 3, 6, 9, and 12
Description: WPAI-SHP is a 6-question participant-rated questionnaire to determine degree to which a specific health problem affected work productivity while at work and outside of work. Four scores are derived: percentage of absenteeism (percentage of work time missed) and presenteeism (reduced productivity while at work), overall work impairment score combining absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. Score range: 0 (not affected/no impairment) to 100 (completely affected/impaired). WPAI outcomes are expressed as impairment percentages with higher numbers indicating greater impairment and less productivity. A decrease from Baseline indicates improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of work time missed
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 191 | 14
percentage of work time missed
  Overall | -2.5 (1.87) | -8.3 (4.60)
  Month 3 | -3.0 (2.15) | -4.0 (5.81)
  Month 6 | -5.3 (1.95) | -7.6 (5.07)
  Month 9 | -1.1 (2.31) | -9.6 (7.77)
  Month 12 | -0.7 (2.24) | -12.1 (6.54)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1795, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0715, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2065, mixed effect model; least squares mean = 5.8, Standard Error of Mean 4.60
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1649, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4894, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8611, mixed effect model; least squares mean = 1.0, Standard Error of Mean 5.89
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0073, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1343, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6468, mixed effect model; least squares mean = 2.3, Standard Error of Mean 5.09
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6441, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2176, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2814, mixed effect model; least squares mean = 8.5, Standard Error of Mean 7.91
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7533, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0653, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage of work time missed due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0876, mixed effect model; least squares mean = 11.4, Standard Error of Mean 6.65

10. Secondary Outcome: Change From Baseline in Percent Impairment While Working Due to MS, by the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of impairment while working
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 217 | 16
percentage of impairment while working
  Overall | -4.2 (1.88) | -8.4 (4.56)
  Month 3 | -6.9 (2.09) | -1.8 (5.53)
  Month 6 | -6.5 (2.01) | -5.6 (5.38)
  Month 9 | -3.0 (2.18) | -17.9 (6.80)
  Month 12 | -0.3 (2.22) | -8.4 (6.80)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0281, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0654, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3400, mixed effect model; least squares mean = 4.3, Standard Error of Mean 4.47
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0012, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7490, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3592, mixed effect model; least squares mean = -5.1, Standard Error of Mean 5.53
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0015, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2967, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8735, mixed effect model; least squares mean = -0.9, Standard Error of Mean 5.34
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1696, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0089, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0297, mixed effect model; least squares mean = 14.9, Standard Error of Mean 6.83
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8806, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2170, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage impairment while working due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2392, mixed effect model; least squares mean = 8.1, Standard Error of Mean 6.86

11. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment Due to MS, by the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of overall work impairment
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 186 | 13
percentage of overall work impairment
  Overall | -5.2 (2.24) | -8.7 (5.69)
  Month 3 | -7.7 (2.49) | -4.5 (6.57)
  Month 6 | -7.8 (2.43) | -2.9 (6.73)
  Month 9 | -2.4 (2.86) | -15.9 (9.83)
  Month 12 | -2.9 (2.47) | -11.7 (7.06)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0219, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1259, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5312, mixed effect model; least squares mean = 3.6, Standard Error of Mean 5.68
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0022, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4968, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6283, mixed effect model; least squares mean = -3.2, Standard Error of Mean 6.64
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0016, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6631, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4770, mixed effect model; least squares mean = -4.8, Standard Error of Mean 6.77
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4027, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1077, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1781, mixed effect model; least squares mean = 13.5, Standard Error of Mean 9.98
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2422, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0994, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of percentage overall work impairment due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2194, mixed effect model; least squares mean = 8.8, Standard Error of Mean 7.13

12. Secondary Outcome: Change From Baseline in Regular Activity Productivity Loss, by the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of activity impairment
Arm/Group | Responder | Non-responder
Number analyzed (Participants) | 650 | 77
percentage of activity impairment
  Overall | -11.4 (1.31) | -4.1 (2.37)
  Month 3 | -13.5 (1.42) | -3.1 (2.83)
  Month 6 | -12.3 (1.43) | -4.7 (2.94)
  Month 9 | -10.4 (1.44) | -4.1 (3.08)
  Month 12 | -9.2 (1.45) | -4.4 (3.20)
Statistical Analysis 1: Comparison: Responder; Overall, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder; Overall, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0860, mixed effect model
Statistical Analysis 3: Comparison: Responder vs Non-responder; Overall, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0010, mixed effect model; least squares mean = -7.3, Standard Error of Mean 2.20
Statistical Analysis 4: Comparison: Responder; Month 3, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Non-responder; Month 3, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2777, mixed effect model
Statistical Analysis 6: Comparison: Responder vs Non-responder; Month 3, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0002, mixed effect model; least squares mean = -10.4, Standard Error of Mean 2.76
Statistical Analysis 7: Comparison: Responder; Month 6, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder; Month 6, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1078, mixed effect model
Statistical Analysis 9: Comparison: Responder vs Non-responder; Month 6, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0082, mixed effect model; least squares mean = -7.6, Standard Error of Mean 2.87
Statistical Analysis 10: Comparison: Responder; Month 9, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Non-responder; Month 9, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1838, mixed effect model
Statistical Analysis 12: Comparison: Responder vs Non-responder; Month 9, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0364, mixed effect model; least squares mean = -6.3, Standard Error of Mean 3.02
Statistical Analysis 13: Comparison: Responder; Month 12, Responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder; Month 12, Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1714, mixed effect model
Statistical Analysis 15: Comparison: Responder vs Non-responder; Month 12, Responder versus Non-responder: Mixed effect model for repeated measures with visit, responder group, visit and responder group interaction, baseline of regular activity productivity loss due to MS, baseline EDSS score, MS disease type, age, gender, total number of relapses experienced within the past 12 months and country as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1259, mixed effect model; least squares mean = -4.8, Standard Error of Mean 3.14

13. Secondary Outcome: Change From Baseline in the PCS of the SF-36 at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the MCS score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Increases from baseline indicate improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Relapsing-Remitting MS: Participants in the Responder group with relapsing-remitting MS (RRMS).
  Participants took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment responders continued 10 mg fampridine twice daily for 44 weeks.
- Secondary-Progressive MS: Participants in the Responder group with secondary-progressive MS (SPMS).
  Participants took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment responders continued 10 mg fampridine twice daily for 44 weeks.
- Primary-Progressive MS: Participants in the Responder group with primary-progressive MS (PPMS).
  Participants took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment responders continued 10 mg fampridine twice daily for 44 weeks.
- Progressive-Relapsing MS: Participants in the Responder group with progressive-relapsing MS (PRMS).
  Participants took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment responders continued 10 mg fampridine twice daily for 44 weeks.
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 256 | 264 | 115 | 31
units on a scale
  Overall | 4.5 (0.39) | 3.8 (0.38) | 2.5 (0.49) | 3.2 (0.89)
  Month 3 | 5.5 (0.42) | 4.5 (0.41) | 3.1 (0.55) | 2.7 (1.01)
  Month 6 | 4.4 (0.46) | 3.9 (0.45) | 2.3 (0.61) | 3.9 (1.13)
  Month 9 | 4.2 (0.45) | 3.2 (0.45) | 3.0 (0.60) | 3.2 (1.12)
  Month 12 | 4.0 (0.45) | 3.4 (0.45) | 1.7 (0.61) | 2.9 (1.14)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0004, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0069, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0001, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0006, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0040, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0047, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline PCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0118, mixed effect model

14. Secondary Outcome: Change From Baseline in the MCS of the SF-36 at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: as for outcome 13
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 256 | 264 | 116 | 31
units on a scale
  Overall | 4.0 (0.59) | 3.0 (0.58) | 3.2 (0.74) | 2.0 (1.36)
  Month 3 | 4.9 (0.64) | 4.5 (0.63) | 3.9 (0.83) | 2.6 (1.54)
  Month 6 | 4.3 (0.67) | 2.9 (0.66) | 3.5 (0.89) | 2.9 (1.65)
  Month 9 | 3.1 (0.70) | 2.1 (0.69) | 2.7 (0.93) | 2.0 (1.74)
  Month 12 | 3.5 (0.68) | 2.6 (0.67) | 2.5 (0.89) | 0.5 (1.68)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.1398, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0935, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0760, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0019, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0037, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.2489, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0001, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0052, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline MCS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.7714, mixed effect model

15. Secondary Outcome: Change From Baseline in the MSIS-29 Physical Score at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: The MSIS-29 is a disease-specific patient-reported outcome measure that has been developed and validated to examine the physical and psychological impact of MS from a patient's perspective; it measures 20 physical items and 9 psychological items. Sum of 20 physical condition items converted into a 0-100 score range, where missing items are imputed by average of total of non-missing items when no more than 50% are missing (otherwise the total score is missing). A lower total score indicates less physically-related impact while a higher total score indicates greater physically-related impact on a participant's functioning. Decreases from Baseline indicate improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 256 | 264 | 118 | 31
units on a scale
  Overall | -12.1 (1.12) | -10.3 (1.09) | -8.3 (1.40) | -12.5 (2.58)
  Month 3 | -15.0 (1.16) | -13.3 (1.13) | -10.6 (1.47) | -12.6 (2.72)
  Month 6 | -12.0 (1.22) | -10.9 (1.19) | -8.4 (1.58) | -14.9 (2.94)
  Month 9 | -10.5 (1.27) | -8.9 (1.25) | -7.9 (1.67) | -10.4 (3.13)
  Month 12 | -10.9 (1.27) | -8.2 (1.25) | -6.2 (1.66) | -11.9 (3.15)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0009, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0002, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 physical score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0002, mixed effect model

16. Secondary Outcome: Change From Baseline in the MSIS-29 Psychological Score at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: The MSIS-29 is a disease-specific patient-reported outcome measure that has been developed and validated to examine the physical and psychological impact of MS from a patient's perspective; it measures 20 physical items and 9 psychological items. Sum of 9 psychological condition items converted into a 0-100 score range, where missing items are imputed by average of total of non-missing items when no more than 50% are missing (otherwise the total score is missing). A lower total score indicates less psychologically-related impact while a higher total score indicates greater psychologically-related impact on a participant's functioning. Decreases from Baseline indicate improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 257 | 263 | 118 | 31
units on a scale
  Overall | -9.4 (1.09) | -6.5 (1.07) | -8.3 (1.37) | -7.5 (2.53)
  Month 3 | -11.2 (1.17) | -8.9 (1.15) | -9.1 (1.51) | -8.6 (2.80)
  Month 6 | -8.8 (1.23) | -6.8 (1.22) | -8.7 (1.62) | -7.9 (3.06)
  Month 9 | -8.3 (1.29) | -5.1 (1.27) | -8.2 (1.70) | -8.3 (3.21)
  Month 12 | -9.3 (1.29) | -5.3 (1.28) | -7.4 (1.71) | -5.1 (3.29)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0032, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0021, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0097, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0103, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline MSIS-29 psychological score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.1227, mixed effect model

17. Secondary Outcome: Change From Baseline in the Activity Limitation Scale (ALS) of PRIMUS Score at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: as for outcome 6
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 198 | 187 | 87 | 26
units on a scale
  Overall | -2.5 (0.29) | -1.1 (0.27) | -0.5 (0.39) | -1.7 (0.70)
  Month 3 | -3.2 (0.31) | -2.1 (0.29) | -1.6 (0.42) | -1.9 (0.77)
  Month 6 | -2.3 (0.35) | -1.3 (0.34) | -0.8 (0.48) | -1.6 (0.88)
  Month 9 | -2.4 (0.35) | -0.7 (0.33) | -0.3 (0.48) | -2.0 (0.88)
  Month 12 | -2.0 (0.37) | -0.5 (0.36) | 0.7 (0.52) | -1.2 (0.97)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1754, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0192, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0157, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0002, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1012, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0749, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0455, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4699, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0235, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1978, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1977, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline of the total ALS score, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2250, mixed effect model

18. Secondary Outcome: Change From Baseline in Current Health State of the EQ-5D VAS at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: as for outcome 7
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 256 | 258 | 116 | 29
units on a scale
  Overall | 8.8 (1.06) | 6.5 (1.04) | 6.7 (1.34) | 4.7 (2.53)
  Month 3 | 10.1 (1.17) | 8.2 (1.15) | 7.3 (1.53) | 4.6 (2.91)
  Month 6 | 8.0 (1.22) | 6.1 (1.21) | 6.0 (1.63) | 4.1 (3.12)
  Month 9 | 8.2 (1.25) | 5.6 (1.24) | 7.9 (1.66) | 5.5 (3.22)
  Month 12 | 8.8 (1.26) | 6.1 (1.26) | 5.5 (1.70) | 4.5 (3.36)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0649, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1138, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0003, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1850, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0887, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0011, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline of the current health state of EQ-5D scores, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1853, mixed effect model

19. Secondary Outcome: Change From Baseline in EQ-5D Index Scores at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: EQ-5D is a participant-answered questionnaire containing a descriptive system on 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression and a VAS on health state. The scores on the 5 dimensions of descriptive system can be converted into an index score by applying UK weights. EQ-5D index score ranges from 1 to -0.59, and 1 reflects the best outcome. An increase from baseline indicates improvement. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error. The 'overall' estimate is the average change from baseline over the whole time period (through Month 12).
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 254 | 262 | 114 | 31
units on a scale
  Overall | 0.05 (0.01) | 0.04 (0.01) | 0.05 (0.02) | 0.07 (0.03)
  Month 3 | 0.07 (0.01) | 0.06 (0.01) | 0.05 (0.02) | 0.06 (0.03)
  Month 6 | 0.04 (0.01) | 0.05 (0.01) | 0.05 (0.02) | 0.09 (0.04)
  Month 9 | 0.05 (0.01) | 0.02 (0.01) | 0.04 (0.02) | 0.02 (0.04)
  Month 12 | 0.04 (0.01) | 0.03 (0.01) | 0.05 (0.02) | 0.10 (0.04)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; p = 0.0005, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; [analysis description as in outcome 18, analysis 3]; Test type: Superiority or Other; p = 0.0027, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.0167, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; [analysis description as in outcome 18, analysis 5]; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; [analysis description as in outcome 18, analysis 6]; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; [analysis description as in outcome 18, analysis 7]; Test type: Superiority or Other; p = 0.0024, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; [analysis description as in outcome 18, analysis 8]; Test type: Superiority or Other; p = 0.0669, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; [analysis description as in outcome 18, analysis 9]; Test type: Superiority or Other; p = 0.0018, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; [analysis description as in outcome 18, analysis 10]; Test type: Superiority or Other; p = 0.0004, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; [analysis description as in outcome 18, analysis 11]; Test type: Superiority or Other; p = 0.0190, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; [analysis description as in outcome 18, analysis 12]; Test type: Superiority or Other; p = 0.0106, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; [analysis description as in outcome 18, analysis 13]; Test type: Superiority or Other; p = 0.0009, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; [analysis description as in outcome 18, analysis 14]; Test type: Superiority or Other; p = 0.1937, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; [analysis description as in outcome 18, analysis 15]; Test type: Superiority or Other; p = 0.0445, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; [analysis description as in outcome 18, analysis 16]; Test type: Superiority or Other; p = 0.6475, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; [analysis description as in outcome 18, analysis 17]; Test type: Superiority or Other; p = 0.0097, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; [analysis description as in outcome 18, analysis 18]; Test type: Superiority or Other; p = 0.0386, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; [analysis description as in outcome 18, analysis 19]; Test type: Superiority or Other; p = 0.0219, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; [analysis description as in outcome 18, analysis 20]; Test type: Superiority or Other; p = 0.0076, mixed effect model

20. Secondary Outcome: Change From Baseline in Percent Work Time Missed Due to MS on the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of work time missed
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 93 | 55 | 34 | 9
percentage of work time missed
  Overall | -2.9 (2.01) | -1.5 (2.51) | -2.5 (2.86) | -4.0 (5.82)
  Month 3 | -3.1 (2.49) | -2.6 (3.18) | -3.3 (3.81) | -1.1 (8.51)
  Month 6 | -6.4 (2.23) | -5.3 (2.79) | -3.3 (3.15) | -2.3 (6.29)
  Month 9 | -1.9 (2.86) | 2.0 (3.68) | -1.1 (4.44) | -10.0 (8.77)
  Month 12 | -0.3 (2.67) | -0.1 (3.44) | -2.2 (4.12) | -2.7 (8.24)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.1471, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.5503, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.3854, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.4893, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.2166, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.4149, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.3849, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.8980, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0046, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0594, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.2975, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.7155, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.5070, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.5848, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.8020, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.2540, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.9057, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.9679, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.5875, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of work time missed due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.7440, mixed effect model

21. Secondary Outcome: Change From Baseline in Percent Impairment While Working Due to MS on the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of impairment while working
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 106 | 62 | 40 | 9
percentage of impairment while working
  Overall | -5.8 (1.95) | -4.2 (2.43) | 0.8 (2.78) | -7.3 (5.95)
  Month 3 | -8.6 (2.28) | -8.0 (2.88) | -1.7 (3.38) | -2.9 (7.57)
  Month 6 | -6.7 (2.20) | -8.7 (2.79) | -2.5 (3.26) | -8.3 (6.88)
  Month 9 | -5.0 (2.49) | -1.8 (3.17) | 0.5 (3.85) | -4.9 (8.51)
  Month 12 | -2.9 (2.56) | 1.4 (3.35) | 6.8 (3.95) | -13.1 (8.38)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0032, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0828, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.7756, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.2200, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0002, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0061, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.6258, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.6987, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0025, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0021, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.4385, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.2275, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0446, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.5757, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.8936, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.5675, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.2539, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.6673, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0849, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of impairment while working due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.1187, mixed effect model

22. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment Due to MS on the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of overall work impairment
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 92 | 52 | 33 | 9
percentage of overall work impairment
  Overall | -7.5 (2.41) | -6.8 (3.09) | -0.8 (3.54) | -6.5 (6.97)
  Month 3 | -10.7 (2.74) | -10.4 (3.56) | -1.7 (4.18) | 2.9 (9.51)
  Month 6 | -9.2 (2.81) | -11.9 (3.60) | -3.3 (4.22) | -6.5 (8.10)
  Month 9 | -4.9 (3.49) | -2.6 (4.61) | 1.2 (5.62) | -9.7 (11.15)
  Month 12 | -5.3 (2.84) | -2.1 (3.73) | 0.4 (4.42) | -12.6 (8.31)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0022, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0299, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.8135, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.3526, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0039, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.6924, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.7639, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0013, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0011, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.4340, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.4224, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.1628, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.5666, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; Month 9, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.8315, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.3852, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0652, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.5719, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.9237, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of overall work impairment due to MS, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.1310, mixed effect model

23. Secondary Outcome: Change From Baseline in Regular Activity Productivity Loss on the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12 by MS Disease Type: Responders
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of activity impairment
Arm/Group | Relapsing-Remitting MS | Secondary-Progressive MS | Primary-Progressive MS | Progressive-Relapsing MS
Number analyzed (Participants) | 251 | 252 | 116 | 31
percentage of activity impairment
  Overall | -14.9 (1.49) | -9.8 (1.47) | -7.1 (1.86) | -12.2 (3.39)
  Month 3 | -16.2 (1.74) | -13.4 (1.72) | -8.7 (2.29) | -11.0 (4.28)
  Month 6 | -15.1 (1.76) | -11.1 (1.76) | -9.0 (2.35) | -14.2 (4.35)
  Month 9 | -14.9 (1.79) | -7.5 (1.78) | -7.1 (2.35) | -10.8 (4.46)
  Month 12 | -13.5 (1.79) | -7.1 (1.79) | -3.7 (2.37) | -13.0 (4.51)
Statistical Analysis 1: Comparison: Relapsing-Remitting MS; Overall, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Secondary-Progressive MS; Overall, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 3: Comparison: Primary-Progressive MS; Overall, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Progressive-Relapsing MS; Overall, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0003, mixed effect model
Statistical Analysis 5: Comparison: Relapsing-Remitting MS; Month 3, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 6: Comparison: Secondary-Progressive MS; Month 3, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 7: Comparison: Primary-Progressive MS; Month 3, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0002, mixed effect model
Statistical Analysis 8: Comparison: Progressive-Relapsing MS; Month 3, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0102, mixed effect model
Statistical Analysis 9: Comparison: Relapsing-Remitting MS; Month 6, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Secondary-Progressive MS; Month 6, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 11: Comparison: Primary-Progressive MS; Month 6, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0001, mixed effect model
Statistical Analysis 12: Comparison: Progressive-Relapsing MS; Month 6, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0012, mixed effect model
Statistical Analysis 13: Comparison: Relapsing-Remitting MS; Month 9, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Secondary-Progressive MS; Month 9, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 15: Comparison: Primary-Progressive MS; [analysis description as in outcome 23, analysis 14]; Test type: Superiority or Other; p = 0.0026, mixed effect model
Statistical Analysis 16: Comparison: Progressive-Relapsing MS; Month 9, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0161, mixed effect model
Statistical Analysis 17: Comparison: Relapsing-Remitting MS; Month 12, RRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 18: Comparison: Secondary-Progressive MS; Month 12, SPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 19: Comparison: Primary-Progressive MS; Month 12, PPMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.1151, mixed effect model
Statistical Analysis 20: Comparison: Progressive-Relapsing MS; Month 12, PRMS. Mixed effect model for repeated measures with visit, baseline of percentage of regular activity productivity loss, MS type, age, gender, country, visit and MS type interaction, baseline EDSS score and total number of relapses experienced within the past 12 months as fixed effects. An unstructured covariance was used to model within-participant error; Test type: Superiority or Other; p = 0.0040, mixed effect model

24. Secondary Outcome: Change From Baseline in the PCS of the SF-36 at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 3
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Responder: Taking Additional MS Therapy: Participants (taking additional MS therapy) took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment responders continued 10 mg fampridine twice daily for 44 weeks.
- Non-responder: Taking Additional MS Therapy: Participants (taking additional MS therapy) took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment non-responders continued without treatment by completing quality of life questionnaires.
- Responder: Not Taking Additional MS Therapy: Participants (not taking additional MS therapy) took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment responders continued 10 mg fampridine twice daily for 44 weeks.
- Non-responder: Not Taking Additional MS Therapy: Participants (not taking additional MS therapy) took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment non-responders continued without treatment by completing quality of life questionnaires.
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 521 | 58 | 145 | 23
units on a scale
  Overall | 3.1 (0.36) | -0.3 (0.71) | 3.9 (0.48) | -0.6 (1.08)
  Month 3 | 4.0 (0.38) | 0.1 (0.77) | 4.1 (0.53) | -1.2 (1.19)
  Month 6 | 3.1 (0.40) | 0.6 (0.89) | 3.9 (0.58) | -0.8 (1.35)
  Month 9 | 2.7 (0.40) | -1.2 (0.91) | 4.0 (0.58) | -0.7 (1.46)
  Month 12 | 2.5 (0.40) | -0.8 (0.94) | 3.6 (0.58) | 0.2 (1.44)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6769, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5780, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 3.4, Standard Error of Mean 0.68
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 4.5, Standard Error of Mean 1.10
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8886, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3221, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 3.9, Standard Error of Mean 0.75
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 5.3, Standard Error of Mean 1.23
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4668, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5695, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0058, mixed effect model; difference of LS means = 2.4, Standard Error of Mean 0.88
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0010, mixed effect model; difference of LS means = 4.6, Standard Error of Mean 1.40
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2040, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6306, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non- responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 3.9, Standard Error of Mean 0.90
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0020, mixed effect model; difference of LS means = 4.7, Standard Error of Mean 1.51
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4052, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8626, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0004, mixed effect model; difference of LS means = 3.3, Standard Error of Mean 0.93
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline PCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0263, mixed effect model; difference of LS means = 3.3, Standard Error of Mean 1.49

25. Secondary Outcome: Change From Baseline in the MCS of the SF-36 at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 3
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 522 | 58 | 145 | 23
units on a scale
  Overall | 2.8 (0.56) | -0.1 (1.09) | 3.9 (0.74) | 0.6 (1.64)
  Month 3 | 4.0 (0.59) | -1.3 (1.18) | 4.8 (0.81) | 1.1 (1.82)
  Month 6 | 3.0 (0.60) | 0.2 (1.29) | 4.1 (0.85) | 1.5 (1.96)
  Month 9 | 2.1 (0.62) | 1.3 (1.40) | 2.8 (0.89) | 0.0 (2.24)
  Month 12 | 2.1 (0.61) | -0.7 (1.40) | 3.9 (0.87) | -0.3 (2.15)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8999, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7156, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0050, mixed effect model; difference of LS means = 2.9, Standard Error of Mean 1.03
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0490, mixed effect model; difference of LS means = 3.3, Standard Error of Mean 1.68
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2740, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5556, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 5.2, Standard Error of Mean 1.15
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0476, mixed effect model; difference of LS means = 3.7, Standard Error of Mean 1.88
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8627, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4312, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0305, mixed effect model; difference of LS means = 2.8, Standard Error of Mean 1.27
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2059, mixed effect model; difference of LS means = 2.6, Standard Error of Mean 2.03
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0008, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3685, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0016, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9862, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5561, mixed effect model; difference of LS means = 0.8, Standard Error of Mean 1.38
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2281, mixed effect model; difference of LS means = 2.8, Standard Error of Mean 2.32
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0006, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6004, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9040, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0401, mixed effect model; difference of LS means = 2.8, Standard Error of Mean 1.38
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the 2-way and 3-way interactions among them, baseline MCS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0651, mixed effect model; difference of LS means = 4.1, Standard Error of Mean 2.23

26. Secondary Outcome: Change From Baseline in the MSIS-29 Physical Score at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 4
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 524 | 57 | 145 | 22
units on a scale
  Overall | -9.6 (1.05) | -1.5 (2.03) | -12.2 (1.38) | -3.2 (3.10)
  Month 3 | -12.6 (1.07) | -1.4 (2.08) | -14.0 (1.43) | -4.0 (3.22)
  Month 6 | -10.0 (1.10) | -2.2 (2.28) | -12.2 (1.52) | -5.2 (3.47)
  Month 9 | -8.0 (1.13) | -0.4 (2.48) | -11.8 (1.61) | 0.5 (4.02)
  Month 12 | -7.8 (1.13) | -2.1 (2.57) | -11.1 (1.61) | -4.3 (3.95)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4540, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2949, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = -8.1, Standard Error of Mean 1.93
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0046, mixed effect model; difference of LS means = -9.0, Standard Error of Mean 3.16
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = -12.6, Standard Error of Mean 1.07
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5020, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2157, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = -11.2, Standard Error of Mean 2.00
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0026, mixed effect model; difference of LS means = -10.0, Standard Error of Mean 3.30
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3435, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1357, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0004, mixed effect model; difference of LS means = -7.8, Standard Error of Mean 2.22
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0511, mixed effect model; difference of LS means = -7.0, Standard Error of Mean 3.58
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8703, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9049, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0019, mixed effect model; difference of LS means = -7.6, Standard Error of Mean 2.44
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0033, mixed effect model; difference of LS means = -12.3, Standard Error of Mean 4.15
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4087, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2755, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0251, mixed effect model; difference of LS means = -5.7, Standard Error of Mean 2.52
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 physical score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0989, mixed effect model; difference of LS means = -6.7, Standard Error of Mean 4.08

27. Secondary Outcome: Change From Baseline in MSIS-29 Psychological Score at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 16
Time Frame: Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 525 | 57 | 144 | 22
units on a scale
  Overall | -7.1 (1.02) | -0.3 (2.00) | -9.7 (1.36) | -2.8 (3.06)
  Month 3 | -9.0 (1.07) | 0.2 (2.17) | -11.1 (1.49) | -1.0 (3.39)
  Month 6 | -7.1 (1.10) | -2.6 (2.37) | -9.5 (1.56) | -2.6 (3.60)
  Month 9 | -6.1 (1.13) | -0.2 (2.57) | -8.9 (1.64) | -2.4 (4.22)
  Month 12 | -6.2 (1.13) | 1.3 (2.70) | -9.1 (1.67) | -5.1 (4.16)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8767, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3673, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0004, mixed effect model; difference of LS means = -6.8, Standard Error of Mean 1.91
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0273, mixed effect model; difference of LS means = -6.9, Standard Error of Mean 3.12
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9091, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7718, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = -9.2, Standard Error of Mean 2.11
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0038, mixed effect model; difference of LS means = -10.1, Standard Error of Mean 3.50
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2720, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4767, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0553, mixed effect model; difference of LS means = -4.5, Standard Error of Mean 2.32
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0632, mixed effect model; difference of LS means = -6.9, Standard Error of Mean 3.73
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9398, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5655, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0204, mixed effect model; difference of LS means = -5.9, Standard Error of Mean 2.54
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; [analysis description as in outcome 27, analysis 21]; Test type: Superiority or Other; p = 0.1414, mixed effect model; difference of LS means = -6.4, Standard Error of Mean 4.37
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6279, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2239, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0049, mixed effect model; difference of LS means = -7.5, Standard Error of Mean 2.67
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline MSIS-29 psychological score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3457, mixed effect model; difference of LS means = -4.1, Standard Error of Mean 4.32

28. Secondary Outcome: Change From Baseline in the Activities Limitation Scale of the PRIMUS at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 6
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 395 | 33 | 103 | 12
units on a scale
  Overall | -1.3 (0.24) | 0.8 (0.63) | -1.9 (0.37) | 0.8 (1.11)
  Month 3 | -2.1 (0.25) | -0.5 (0.67) | -2.9 (0.40) | -0.0 (1.14)
  Month 6 | -1.2 (0.27) | 0.6 (0.81) | -2.1 (0.46) | 1.3 (1.33)
  Month 9 | -1.1 (0.27) | 2.0 (0.82) | -1.6 (0.46) | 1.1 (1.67)
  Month 12 | -0.7 (0.29) | 1.1 (0.93) | -1.0 (0.50) | 1.0 (1.81)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2087, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4487, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0013, mixed effect model; difference of LS means = -2.1, Standard Error of Mean 0.64
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0188, mixed effect model; difference of LS means = -2.7, Standard Error of Mean 1.15
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4243, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9989, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0207, mixed effect model; difference of LS means = -1.6, Standard Error of Mean 0.68
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0161, mixed effect model; difference of LS means = -2.9, Standard Error of Mean 1.18
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4256, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3313, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0238, mixed effect model; difference of LS means = -1.9, Standard Error of Mean 0.83
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0150, mixed effect model; difference of LS means = -3.4, Standard Error of Mean 1.39
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0171, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0007, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5146, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0003, mixed effect model; difference of LS means = -3.0, Standard Error of Mean 0.84
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1224, mixed effect model; difference of LS means = -2.7, Standard Error of Mean 1.72
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0168, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2272, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0570, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5832, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0561, mixed effect model; difference of LS means = -1.8, Standard Error of Mean 0.94
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the total ALS score, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2971, mixed effect model; difference of LS means = -1.9, Standard Error of Mean 1.86

29. Secondary Outcome: Change From Baseline in the Current Health State of EQ-5D VAS at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 7
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 518 | 58 | 141 | 21
units on a scale
  Overall | 6.0 (1.00) | -5.8 (1.95) | 8.6 (1.33) | -0.8 (3.04)
  Month 3 | 7.6 (1.06) | -3.9 (2.16) | 8.6 (1.49) | -1.2 (3.46)
  Month 6 | 5.2 (1.09) | -5.6 (2.35) | 8.6 (1.56) | 1.5 (3.72)
  Month 9 | 5.5 (1.11) | -6.1 (2.51) | 8.7 (1.62) | -1.8 (4.13)
  Month 12 | 5.5 (1.12) | -7.7 (2.67) | 8.7 (1.67) | -1.5 (4.33)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0029, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8041, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 11.8, Standard Error of Mean 1.85
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0026, mixed effect model; difference of LS means = 9.4, Standard Error of Mean 3.10
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0689, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7182, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 11.6, Standard Error of Mean 2.10
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0061, mixed effect model; difference of LS means = 9.8, Standard Error of Mean 3.57
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0179, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6911, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 10.8, Standard Error of Mean 2.31
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0666, mixed effect model; difference of LS means = 7.1, Standard Error of Mean 3.85
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0158, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6684, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 11.6, Standard Error of Mean 2.49
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0141, mixed effect model; difference of LS means = 10.5, Standard Error of Mean 4.28
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0042, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7329, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model; difference of LS means = 13.2, Standard Error of Mean 2.65
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0242, mixed effect model; difference of LS means = 10.1, Standard Error of Mean 4.49

30. Secondary Outcome: Change From Baseline in the Index Scores of EQ-5D at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 19
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 519 | 56 | 142 | 22
units on a scale
  Overall | 0.04 (0.01) | -0.00 (0.02) | 0.06 (0.02) | 0.02 (0.03)
  Month 3 | 0.07 (0.01) | 0.02 (0.02) | 0.07 (0.02) | -0.02 (0.04)
  Month 6 | 0.05 (0.01) | -0.00 (0.03) | 0.05 (0.02) | 0.03 (0.04)
  Month 9 | 0.03 (0.01) | -0.00 (0.03) | 0.06 (0.02) | 0.02 (0.05)
  Month 12 | 0.03 (0.01) | -0.03 (0.03) | 0.07 (0.02) | 0.04 (0.05)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9151, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6128, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0331, mixed effect model; difference of LS means = 0.05, Standard Error of Mean 0.02
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1919, mixed effect model; difference of LS means = 0.05, Standard Error of Mean 0.04
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4481, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5454, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0516, mixed effect model; difference of LS means = 0.05, Standard Error of Mean 0.02
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0175, mixed effect model; difference of LS means = 0.09, Standard Error of Mean 0.04
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9371, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0056, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5475, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0699, mixed effect model; difference of LS means = 0.05, Standard Error of Mean 0.03
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5870, mixed effect model; difference of LS means = 0.02, Standard Error of Mean 0.05
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0245, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9926, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0027, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6368, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3358, mixed effect model; difference of LS means = 0.03, Standard Error of Mean 0.03
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5089, mixed effect model; difference of LS means = 0.03, Standard Error of Mean 0.05
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0141, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4280, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0002, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3827, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0748, mixed effect model; difference of LS means = 0.06, Standard Error of Mean 0.03
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the current health state of EQ-5D index scores, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5663, mixed effect model; least squares mean = 0.03, Standard Error of Mean 0.05

31. Secondary Outcome: Change From Baseline in Percent Work Time Missed Due to MS on the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of work time missed
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 149 | 12 | 42 | 2
percentage of work time missed
  Overall | -3.0 (2.10) | -11.9 (4.93) | -2.4 (2.72) | 14.9 (12.11)
  Month 3 | -3.7 (2.43) | -8.3 (6.14) | -2.0 (3.43) | 28.6 (17.71)
  Month 6 | -6.0 (2.21) | -10.3 (5.52) | -4.3 (2.98) | 6.4 (12.11)
  Month 9 | -1.2 (2.60) | -12.8 (8.32) | -2.1 (4.09) | 13.9 (21.98)
  Month 12 | -1.0 (2.53) | -16.2 (7.16) | -1.1 (3.79) | 10.6 (15.59)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1544, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0167, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3868, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2214, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0743, mixed effect model; difference of LS means = 8.9, Standard Error of Mean 4.96
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1601, mixed effect model; difference of LS means = -17.2, Standard Error of Mean 12.22
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1251, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1764, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5528, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; [analysis description as in outcome 31, analysis 8]; Test type: Superiority or Other; p = 0.1080, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4644, mixed effect model; difference of LS means = 4.6, Standard Error of Mean 6.27
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0887, mixed effect model; difference of LS means = -30.6, Standard Error of Mean 17.91
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0071, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0640, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1552, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5979, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4444, mixed effect model; difference of LS means = 4.3, Standard Error of Mean 5.58
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3863, mixed effect model; difference of LS means = -10.7, Standard Error of Mean 12.27
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6352, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1265, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6161, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5280, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1769, mixed effect model; difference of LS means = 11.5, Standard Error of Mean 8.51
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4743, mixed effect model; difference of LS means = -16.0, Standard Error of Mean 22.24
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6901, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0245, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7707, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4989, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0387, mixed effect model; difference of LS means = 15.2, Standard Error of Mean 7.31
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % work time missed due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4635, mixed effect model; difference of LS means = -11.7, Standard Error of Mean 15.88

32. Secondary Outcome: Change From Baseline in Percent Impairment While Working Due to MS on the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of impairment while working
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 168 | 13 | 49 | 3
percentage of impairment while working
  Overall | -3.1 (2.10) | -7.3 (5.00) | -6.4 (2.69) | -11.5 (10.86)
  Month 3 | -6.1 (2.35) | -1.0 (6.02) | -8.1 (3.24) | -3.3 (14.07)
  Month 6 | -5.6 (2.26) | -3.8 (5.89) | -8.0 (3.06) | -15.9 (13.27)
  Month 9 | -1.9 (2.44) | -19.0 (7.31) | -5.6 (3.55) | -6.0 (18.93)
  Month 12 | 1.1 (2.49) | -5.5 (7.56) | -3.8 (3.65) | -20.7 (15.27)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1392, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1448, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0187, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2920, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3968, mixed effect model; difference of LS means = 4.2, Standard Error of Mean 4.95
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6420, mixed effect model; difference of LS means = 5.1, Standard Error of Mean 10.95
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0100, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8634, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0134, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8147, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4035, mixed effect model; difference of LS means = -5.1, Standard Error of Mean 6.06
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7385, mixed effect model; difference of LS means = -4.8, Standard Error of Mean 14.25
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0139, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5207, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0091, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2312, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7578, mixed effect model; difference of LS means = -1.8, Standard Error of Mean 5.89
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5575, mixed effect model; difference of LS means = 7.9, Standard Error of Mean 13.42
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4486, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0102, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1185, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7523, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0214, mixed effect model; difference of LS means = 17.1, Standard Error of Mean 7.38
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9826, mixed effect model; difference of LS means = 0.4, Standard Error of Mean 19.12
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6627, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4674, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2965, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1778, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3903, mixed effect model; difference of LS means = 6.6, Standard Error of Mean 7.65
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % impairment while working due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2794, mixed effect model; difference of LS means = 16.8, Standard Error of Mean 15.53

33. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment Due to MS on the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of overall work impairment
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 145 | 11 | 41 | 2
percentage of overall work impairment
  Overall | -4.8 (2.55) | -9.9 (6.26) | -6.7 (3.32) | 1.2 (14.53)
  Month 3 | -7.9 (2.84) | -6.6 (6.99) | -7.1 (3.85) | 18.0 (21.17)
  Month 6 | -7.8 (2.78) | -1.8 (7.48) | -7.7 (3.85) | -8.2 (15.87)
  Month 9 | -1.6 (3.22) | -18.5 (10.69) | -5.5 (5.15) | 3.7 (25.71)
  Month 12 | -1.8 (2.81) | -12.6 (7.95) | -6.5 (4.02) | -8.6 (15.29)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0628, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1166, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0451, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9327, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4177, mixed effect model; difference of LS means = 5.1, Standard Error of Mean 6.28
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5885, mixed effect model; difference of LS means = -7.9, Standard Error of Mean 14.64
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0059, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3467, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0654, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.3965, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8548, mixed effect model; difference of LS means = -1.3, Standard Error of Mean 7.11
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2405, mixed effect model; difference of LS means = -25.1, Standard Error of Mean 21.35
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0056, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8105, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0470, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6067, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4309, mixed effect model; difference of LS means = -6.0, Standard Error of Mean 7.56
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9761, mixed effect model; difference of LS means = 0.5, Standard Error of Mean 16.09
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.6261, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0860, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2884, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8854, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1226, mixed effect model; difference of LS means = 16.9, Standard Error of Mean 10.88
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7249, mixed effect model; difference of LS means = -9.2, Standard Error of Mean 26.07
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5129, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1138, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1086, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.5746, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1831, mixed effect model; difference of LS means = 10.8, Standard Error of Mean 8.07
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the % overall work impairment due to MS, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.8917, mixed effect model; difference of LS means = 2.1, Standard Error of Mean 15.54

34. Secondary Outcome: Change From Baseline in Regular Activity Productivity Loss on the WPAI-SHP Questionnaire at Months 3, 6, 9, and 12 by Whether Taking Additional MS Therapy
Description: as for outcome 9
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of activity impairment
Arm/Group | Responder: Taking Additional MS Therapy | Non-responder: Taking Additional MS Therapy | Responder: Not Taking Additional MS Therapy | Non-responder: Not Taking Additional MS Therapy
Number analyzed (Participants) | 509 | 56 | 141 | 21
percentage of activity impairment
  Overall | -10.6 (1.39) | -4.2 (2.69) | -13.3 (1.83) | -3.1 (4.15)
  Month 3 | -12.7 (1.53) | -3.4 (3.24) | -15.7 (2.20) | -1.8 (5.15)
  Month 6 | -11.5 (1.54) | -6.3 (3.40) | -14.6 (2.23) | -0.5 (5.20)
  Month 9 | -9.8 (1.55) | -5.9 (3.50) | -12.0 (2.28) | 1.6 (5.86)
  Month 12 | -8.5 (1.56) | -1.3 (3.70) | -10.9 (2.31) | -11.6 (5.72)
Statistical Analysis 1: Comparison: Responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 2: Comparison: Non-responder: Taking Additional MS Therapy; Overall, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1152, mixed effect model
Statistical Analysis 3: Comparison: Responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 4: Comparison: Non-responder: Not Taking Additional MS Therapy; Overall, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.4578, mixed effect model
Statistical Analysis 5: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Overall, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0125, mixed effect model; difference of LS means = -6.4, Standard Error of Mean 2.56
Statistical Analysis 6: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Overall, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0158, mixed effect model; difference of LS means = -10.2, Standard Error of Mean 4.23
Statistical Analysis 7: Comparison: Responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 8: Comparison: Non-responder: Taking Additional MS Therapy; Month 3, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2894, mixed effect model
Statistical Analysis 9: Comparison: Responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 10: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 3, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7230, mixed effect model
Statistical Analysis 11: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 3, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0038, mixed effect model; difference of LS means = -9.3, Standard Error of Mean 3.20
Statistical Analysis 12: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 3, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0097, mixed effect model; difference of LS means = -13.9, Standard Error of Mean 5.37
Statistical Analysis 13: Comparison: Responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 14: Comparison: Non-responder: Taking Additional MS Therapy; Month 6, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0628, mixed effect model
Statistical Analysis 15: Comparison: Responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 16: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 6, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9232, mixed effect model
Statistical Analysis 17: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 6, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.1249, mixed effect model; difference of LS means = -5.2, Standard Error of Mean 3.37
Statistical Analysis 18: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 6, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0093, mixed effect model; difference of LS means = -14.1, Standard Error of Mean 5.42
Statistical Analysis 19: Comparison: Responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 20: Comparison: Non-responder: Taking Additional MS Therapy; Month 9, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0937, mixed effect model
Statistical Analysis 21: Comparison: Responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 22: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 9, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7814, mixed effect model
Statistical Analysis 23: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 9, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.2561, mixed effect model; difference of LS means = -3.9, Standard Error of Mean 3.47
Statistical Analysis 24: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 9, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0255, mixed effect model; difference of LS means = -13.6, Standard Error of Mean 6.07
Statistical Analysis 25: Comparison: Responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 26: Comparison: Non-responder: Taking Additional MS Therapy; Month 12, Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.7241, mixed effect model
Statistical Analysis 27: Comparison: Responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p < 0.0001, mixed effect model
Statistical Analysis 28: Comparison: Non-responder: Not Taking Additional MS Therapy; Month 12, Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0427, mixed effect model
Statistical Analysis 29: Comparison: Responder: Taking Additional MS Therapy vs Non-responder: Taking Additional MS Therapy; Month 12, Responder (Taking Additional MS Therapy) versus Non-responder (Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.0498, mixed effect model; difference of LS means = -7.2, Standard Error of Mean 3.67
Statistical Analysis 30: Comparison: Responder: Not Taking Additional MS Therapy vs Non-responder: Not Taking Additional MS Therapy; Month 12, Responder (Not Taking Additional MS Therapy) versus Non-responder (Not Taking Additional MS Therapy): Mixed effect model for repeated measures with visit, responder group, additional MS therapy, the two-way and three-way interactions among them, baseline of the regular activity productivity loss, age, gender, country, baseline EDSS score and total number of relapses experienced as fixed effects. An unstructured covariance was used to model within-patient error; Test type: Superiority or Other; p = 0.9078, mixed effect model; difference of LS means = 0.7, Standard Error of Mean 5.95

35. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: AE: any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. SAE: any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigator, placed the subject at immediate risk of death (a life threatening event); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, could have jeopardized the subject or may have required intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: From signing of Informed Consent (SAEs) or from first dose of study treatment (AEs) through Week 50 or Early Termination (14 +/- 7 days after last dose)
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- All Participants: All participants took 10 mg fampridine twice daily for the first 4 weeks. Those deemed treatment responders continued 10 mg fampridine twice daily for 44 weeks. Those deemed treatment non-responders continued without treatment by completing quality of life questionnaires.
Arm/Group | Responder | Non-responder | All Participants
Number analyzed (Participants) | 707 | 128 | 835
participants
  AE | 522 | 64 | 586
  SAE | 76 | 3 | 79
  Severe AE | 48 | 2 | 50
  Study treatment related AE | 248 | 37 | 285
  Study treatment related SAE | 7 | 0 | 7
  Death | 2 | 0 | 2
  AE leading to study drug discontinuation | 32 | 8 | 40
  AE leading to study discontinuation | 18 | 1 | 19

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent (SAEs) or from first dose of study treatment (AEs) through Week 50 or Early Termination (14 +/- 7 days after last dose).
Arm/Group | Responder | Non-responder | All Participants
Serious Adverse Events (participants affected / at risk) | 76/707 | 3/128 | 79/835
Other Adverse Events (participants affected / at risk) | 314/707 | 41/128 | 355/835
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Responder (N=707) | Non-responder (N=128) | All Participants (N=835)
Multiple Sclerosis Relapse (Nervous system disorders) | 19 | 0 | 19
Grand Mal Convulsion (Nervous system disorders) | 2 | 0 | 2
Multiple Sclerosis (Nervous system disorders) | 2 | 0 | 2
Cerebral Venous Thrombosis (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Muscle Spasticity (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0 | 1
Progressive Multiple Sclerosis (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Trigeminal Neuralgia (Nervous system disorders) | 1 | 0 | 1
Uhthoff's Phenomenon (Nervous system disorders) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 9 | 0 | 9
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Avulsion Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 4
Appendicitis (Infections and infestations) | 1 | 0 | 1
Chronic Sinusitis (Infections and infestations) | 1 | 0 | 1
Gastrointestinal Viral Infection (Infections and infestations) | 1 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 1
Pneumonia Influenzal (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiovascular Disorder (Cardiac disorders) | 1 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Malignant Melanoma Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Hypomania (Psychiatric disorders) | 1 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 1
Bladder Disorder (Renal and urinary disorders) | 1 | 0 | 1
Bladder Dysfunction (Renal and urinary disorders) | 1 | 0 | 1
Liposuction (Surgical and medical procedures) | 1 | 0 | 1
Stent Placement (Surgical and medical procedures) | 1 | 0 | 1
Stent Removal (Surgical and medical procedures) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Death (General disorders) | 1 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 1
Fluid Retention (Metabolism and nutrition disorders) | 0 | 1 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Responder (N=707) | Non-responder (N=128) | All Participants (N=835)
Headache (Nervous system disorders) | 74 | 6 | 80
Multiple Sclerosis Relapse (Nervous system disorders) | 63 | 2 | 65
Dizziness (Nervous system disorders) | 35 | 8 | 43
Urinary Tract Infection (Infections and infestations) | 58 | 7 | 65
Nasopharyngitis (Infections and infestations) | 60 | 1 | 61
Nausea (Gastrointestinal disorders) | 60 | 6 | 66
Insomnia (Psychiatric disorders) | 83 | 12 | 95
Fatigue (General disorders) | 31 | 7 | 38
Fall (Injury, poisoning and procedural complications) | 50 | 5 | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.